CLINICAL TRIAL: NCT04330313
Title: Use of Different Electrophysical Agents in Cervical Region Flexibility Training of Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, ATİYE KAŞ ÖZDEMİR, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018KRM019
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Cervical Flexibility; Stretch; Physical Therapy; Electrotherapy
Keywords: exercise; hotpack; laser therapy; traction
MeSH Terms: conditions — Motor Activity | interventions — Traction; Laser Therapy

STUDY DESIGN:
Intervention Model Description: There are paralel groups, each has 15 participants. Different electrotherapy applications will be applied to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traction and stretching (Experimental): This grup received stretching exercises after traction therapy for 18 sessions, 3 times per week.
  Interventions: Procedure: Traction; Procedure: Stretching
- Laser therapy and stretching (Experimental): This grup received stretching exercises after laser therapy for 18 sessions, 3 times per week.
  Interventions: Procedure: Laser therapy; Procedure: Stretching
- Hot pack and stretching (Experimental): This grup received stretching exercises after hotpack therapy for 18 sessions, 3 times per week.
  Interventions: Procedure: Hot pack; Procedure: Stretching
- Stretching only (Experimental): This grup received only stretching exercises for 18 sessions, 3 times per week.
  Interventions: Procedure: Stretching

INTERVENTIONS:
Procedure: Traction — Intermittent traction will be applied to the cervical region in a supine position with the neck at 25-30 ° flexion. The target weight is determined as 10% of the patient's weight. Traction pulling force applied to the target weight will be achieved gradually increasing from low. Traction therapy will be applied intermittent traction for 15 minutes in each session as 60 seconds retention and 60 seconds rest. The therapy will be held for 18 sessions, 3 days / week.
  Arms: Traction and stretching
Procedure: Laser therapy — Laser therapy will be applied to the participants with a GaAs laser with 904 nm wavelength, 6 points transforaminally, 120 seconds to each point, at 2 J / cm² density, total dose of 12 J laser therapy by keeping the probe in constant contact with the skin.
  Arms: Laser therapy and stretching
Procedure: Hot pack — The hot pack, which is the superficial heat agent, will be held in the neck area of the participants for 20 minutes in each session.The therapy will be held for 18 sessions, 3 days / week.
  Arms: Hot pack and stretching
Procedure: Stretching — Stretching exercises will be repeated 3 times a day in total, 2 times a day self-stretching at home and 1 time under the supervision of a physiotherapist. Exercises for upper trapezius muscle, sternokleudomasteudeus (SCM) muscle and the scalene muscle to be applied in a 3 repeat by waiting 30 seconds, stretching under tension.The therapy will be held for 18 sessions, 3 days / week.

SUMMARY:
60 healthy participants with right / left upper trapezoidal shortness based on volunteering will be included in the study. Participants were randomly divided into 4 groups; Traction and stretching exercises to group 1 (n = 15), laser therapy and stretching exercise to group 2 (n = 15), hot pack and stretching exercises to group 3 (n = 15), and group 4 (control group) only stretching exercises will be applied.

DETAILED DESCRIPTION:
Healthy individuals without any cervical region pathology will be included in the study. Exclusion criterias are pregnancy or cancer, hypertension that cannot be controlled, having neurological symptoms, previous spinal surgery.

Demographic information of the participants will be recorded; cervical joint range of motion (CROM device), muscle shortness (acromion-earlobe and occiput-wall distance measurement), deep cervical flexor muscle strength (Stabilizer Pressure Biofeedback), cervical performance level (Cervical Performance Tests), muscle spasm (Palpable Muscle Spasm Scoring) will be evaluated. Cervical joint range of motion and muscle shortening will be repeated before and after each session, but other parameters will only be repeated at the beginning and the end.

ELIGIBILITY:
Inclusion Criteria:

-Healthy individuals without any cervical region pathology

Exclusion Criteria:

* Pregnancy and cancer
* Uncontrolled hypertension
* Presence of neurological symptoms
* Spinal surgery history

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Cervical range of motion (ROM) | Baseline to 6 weeks after
  ROM is measured by CROM device during flexion, extension, right/left lateral flexion and right/left rotation activity.
Cervical flexibility | Baseline to 6 weeks after
  Cervical flexibility is measured using the standard tape measure, the distance between the occiput and the wall in the standing position of the participants, and the distance between the earlobe and the acromion.

SECONDARY OUTCOMES:
Cervikal Muscle spasm | Baseline to 6 weeks after
  The degree of muscular spasm in the upper trapezoidal muscle, sternocleudomasteudeus (SCM) muscle, and scalen muscles is evaluated by palpation over 4 points.

OTHER OUTCOMES:
Cervical Performance Level | Baseline to 6 weeks after
  In cervical flexion, extension, right and left lateral flexion directions, cervical performance tests are evaluated by recording the holding time in the desired position with a stopwatch.
Muscle Strength of Deep Cervical Flexor Muscles | Baseline to 6 weeks after
  Strength measurement of deep cervical flexor muscles is evaluated with the Stabilizer Pressure Biofeedback device (Chattanooga Medical Suplly Inc, Chattanooga, TN).

CONTACTS AND LOCATIONS:
Overall Officials: Şule ŞİMŞEK, PhD, Study Chair — Pamukkale University; Ummuhan BAŞ ASLAN, Prof. Dr., Study Chair — Pamukkale University; Merve BERGİN KORKMAZ, Dr., Study Chair — Denizli Devlet Hastanesi
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no web site to share data

REFERENCES:
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Hudswell, S., von Mengersen, M., Lucas, N. The cranio-cervical flexion test using pressure biofeedback: A useful measure of cervical dysfunction in the clinical setting? International Journal of Osteopathic Medicine. 2005; 8(3): 98-105.
- [Background] Shahidi B, Johnson CL, Curran-Everett D, Maluf KS. Reliability and group differences in quantitative cervicothoracic measures among individuals with and without chronic neck pain. BMC Musculoskelet Disord. 2012 Oct 31;13:215. doi: 10.1186/1471-2474-13-215. PMID 23114092
- [Background] Zhang LL, Zhou GQ, Qi ZY, He XJ, Li JX, Tang LL, Mao YP, Lin AH, Ma J, Sun Y. Patient- and treatment-related risk factors associated with neck muscle spasm in nasopharyngeal carcinoma patients after intensity-modulated radiotherapy. BMC Cancer. 2017 Nov 23;17(1):788. doi: 10.1186/s12885-017-3780-9. PMID 29169335